CLINICAL TRIAL: NCT04238884
Title: Randomized and Multicenter Clinical Trial to Evaluate the Effectiveness and Efficiency of a Voriconazole Preemptive Genotyping Strategy in Patients With Risk of Aspergillosis
Brief Title: Effectiveness and Efficiency of a Voriconazole Preemptive Genotyping Strategy
Acronym: VORIGENPHARM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-000376-41
Record Dates: First submitted 2020-01-18; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Invasive Fungal Infections
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Based on the genetic study carried out and the patient's characteristics (age, weight, indication), the Pharmacogenetics Unit of the University Hospital La Paz will indicate the dose to be administered based on the therapeutic individualization protocol guided by pharmacogenetics.
  Interventions: Drug: Voriconazole preemptive genotyping strategy
- Control group (Active Comparator): No information will be provided and procedure will be carried out according to normal clinical practice, with clinical monitoring by the doctor in charge.
  Interventions: Drug: Voriconazole clinical practice

INTERVENTIONS:
Drug: Voriconazole preemptive genotyping strategy — The patients who finally receives voriconazole will be randomized to receive the dose according to a pharmacogenetic algorithm including CYP2C19 genotype and clinical and demographic information.
  Arms: Experimental group
Drug: Voriconazole clinical practice — The patients who finally receives voriconazole will be randomized to receive the dose according to clinical practice
  Arms: Control group

SUMMARY:
This is a phase IV pragmatic, multicentre, randomised, simple-blind, parallel arm, centre-stratified clinical trial. The main objective is to compare efficiency of voriconazole preemptive genotyping strategy, compared with routine practice.

DETAILED DESCRIPTION:
Primary outcome is serum level of voriconazole on fifth day. Secondary outcome is a combined variable of therapeutic failure and adverse events, associated with voriconazole. A total of 146 patients with risk of undergoing invasive aspergillosis who potentially will receive voriconazole will be recruited, and CYP2C19 will be genotyped. If the patient receives voriconazole finally, he will be randomized (1:1 experimental/control). In the experimental arm patients receive dose according to pharmacogenetic algorithm including CYP2C19 genotype and clinical and demographic information. In the control arm patients receive dose according to clinical practice guidelines. In addition, a Spain national health system (NHS) point-of-view cost-effectiveness evaluation is going to be done. Direct costs calculation of each arm will be done.

ELIGIBILITY:
Inclusion Criteria:

1. Patient at risk of developing invasive aspergillosis, that will potentially receive treatment or prophylaxis with voriconazole:

   A. Pediatric population: children who are going to receive a transplant of hematopoietic precursors (HSCT) and acute myeloid leukemias, as well as relapses of it.

   B. Adult population: patients diagnosed with acute leukemia, and those patients with expected prolonged neutropenia, secondary to hematological process and / or after specific treatment (aplastic anemia and variants, myelodysplastic syndrome, solid organ or bone marrow transplant, etc.), and those whose responsible clinician consider individually that they could present a risk of developing a fungal infection.
2. Those who agree to participate in the study by signing informed consent (patients equal or over 18 years old)
3. Subjects under 18 years old whose representative / legal guardian has voluntarily signed the informed consent.
4. In the case of mature under 18 years subjects (12-17 years of age), in addition to the consent signed by the legal guardian, the consent of the subject will be obtained.

Exclusion Criteria:

1. Patients who for any reason should not be included in the study according to the criteria of the research team.
2. Subjects who are not capable to understand the information sheet and unable to sign the informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-01-18 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum voriconazole concentration | Day 5 of treatment
  Serum voriconazole concentration within the therapeutic range, in μg/mL.

SECONDARY OUTCOMES:
Therapeutic failure | Within 3 months
  % of patients with therapeutic failure. A patient has a therapeutic failure if:
  1. In patient with suspected or confirmed invasive aspergillosis: drug change or association, because of bad clinical or radiological evolution of the disease.
  2. In patient who receive prophylactic treatment: the necessity of change because of suspected or confirmed invasive fungal disease.
Adverse event | Within 3 months
  % of patients with a dose-dependent drug adverse event reaction.
  It will be considered dose-dependent drug adverse reactions:
  * Visual disturbances (photopsias)
  * Skin reactions
  * Neurotoxicity (confusion and visual hallucinations) and
  * Corrected QT interval (QTc) lengthening
Costs by adverse event | Day 90 of treatment
  Quantifying economic burden (in euros) associated with management of severe adverse events.
Quality adjusted life years (QALY) | Day 90 of treatment
  Measure of disease burden, including both the quality and the quantity of life lived.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto M Borobia, MD, PhD, Principal Investigator — La Paz University Hospital
Locations (1):
- La Paz University Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Monserrat Villatoro J, Garcia Garcia I, Bueno D, de la Camara R, Estebanez M, Lopez de la Guia A, Abad-Santos F, Anton C, Mejia G, Otero MJ, Ramirez Garcia E, Frias Iniesta J, Carcas A, Borobia AM. Randomised multicentre clinical trial to evaluate voriconazole pre-emptive genotyping strategy in patients with risk of aspergillosis: vorigenipharm study protocol. BMJ Open. 2020 Oct 1;10(10):e037443. doi: 10.1136/bmjopen-2020-037443. PMID 33004392